CLINICAL TRIAL: NCT00505505
Title: Effects of Intensive Insulin Therapy on Mortality, Morbidity and Long Term Neurologic Outcome in Neurosurgical Intensive Care Patients
Brief Title: Intensive Insulin Therapy for Strict Glycemic Control in Neurosurgical Patients: Safety and Efficacy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1781964
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2007-07

CONDITIONS: Subarachnoid Hemorrhage; Traumatic Brain Injury; Intracranial Hemorrhage
Keywords: Neurointensive care; Intensive insulin infusion; Hypoglycemia; Postoperative Mortality; Postoperative Morbidity; Neurologic outcome
MeSH Terms: conditions — Subarachnoid Hemorrhage; Brain Injuries, Traumatic; Intracranial Hemorrhages; Hypoglycemia | interventions — insulin, neutral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Insulin infusion rate titrated to maintain glycemia between 80 and 100 mg/dl
  Interventions: Drug: Insulin (Actrapid)
- B (Active Comparator): Insulin infusion rate titrated to maintain glycemia between 80 and 220 mg/dl
  Interventions: Drug: Insulin (Actrapid)

INTERVENTIONS:
Drug: Insulin (Actrapid) — 50 UI Actrapid diluted in 50 ml of saline

SUMMARY:
Strict glycemic control improves mortality and morbidity of patients admitted to the postoperative intensive care unit (ICU). The investigators would like to know if this therapy could improve the long term neurologic and cognitive outcomes of patients treated for acute subarachnoid hemorrhage with either a surgical or intravascular approach.

DETAILED DESCRIPTION:
Intensive Insulin Therapy and Strict Glycemic Control (80-120 mg/dL) Versus Standard Insulin Therapy in Neurosurgical Intensive Care Patients (Subarachnoid Hemorrhage, Traumatic Brain Injury, Intracranial Expanding Lesion): Safety, and Efficacy (Mortality, Morbidity, Long Term Neurologic Outcome).

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage
* Traumatic brain injury
* Intracranial hemorrhage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2002-01

PRIMARY OUTCOMES:
Episodes of hypoglycemia

SECONDARY OUTCOMES:
Infection rate | during the study
Vasospasm rate | during the study
Mortality | 6 months follow up
Neurologic status | 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Federico Bilotta, MD, PhD, Study Chair — Department of Anesthesiology, Critical Care and Pain Medicine
Locations (1):
- University of Rome La Sapienza, Rome, Italy